CLINICAL TRIAL: NCT01170390
Title: Improving Contraceptive Effectiveness in Obese Women
Brief Title: Oral Contraceptives and Body Mass Index
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Alison Edelman, Associate Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: OHSU FAMPLAN 5382; R01HD061582 (NIH)
Record Dates: First submitted 2009-10-27; First posted 2010-07-27 (Estimated); Results first posted 2015-11-26 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-11

CONDITIONS: Body Weight; Contraceptive Usage
Keywords: Obesity; Body weight; Oral contraception; Efficacy
MeSH Terms: conditions — Body Weight; Contraception Behavior; Obesity | interventions — ethinyl estradiol, levonorgestrel drug combination; Ethinyl Estradiol-Norgestrel Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- All participants (Other): A low dose oral contraceptive given cyclically (21 days of active pills/cycle with a 7 day hormonal-free interval) for 2 cycles (56 days).
  Interventions: Drug: All participants (Aviane)
- Aviane and Portia (Active Comparator): A low dose oral contraceptive given cyclically (30mcg EE component, 21 days of active pills/cycle with a 7 day hormonal-free interval) for two cycles
  Interventions: Drug: Portia
- Aviane & Aviane (Active Comparator): A very-low dose oral contraceptive given continuously for 56 days (20mcg EE component, 28 days of active pills/cycle with no hormone free interval)
  Interventions: Drug: Aviane

INTERVENTIONS:
Drug: All participants (Aviane) — 20 mcg EE/0.1 mg LNG cyclically
  Other Names: Levonorgestrel and Ethinyl Estradiol
  Arms: All participants
Drug: Portia — 30 mcg EE/0.15 mg LNG cyclically
  Other Names: Levonorgestrel and Ethinyl Estradiol
  Arms: Aviane and Portia
Drug: Aviane — 20 mcg EE/0.1 mg LNG continuously dosed
  Other Names: Levonorgestrel and Ethinyl Estradiol
  Arms: Aviane & Aviane

SUMMARY:
The main hypothesis for this study is that increased Body Mass Index (BMI) alters oral contraceptive metabolism in a manner which results in decreased effectiveness in obese women.

DETAILED DESCRIPTION:
This study is being conducted to understand how effective oral hormonal birth control (the pill) is for women with high body mass index ("BMI" - the ratio of your height and weight BMI"). Previous studies of birth control traditionally do not include women above a certain BMI number, so safety and efficacy is not clearly understood in this population, yet the pill is still widely used in women with high BMI.

Reproductive-aged, ovulatory women of obese (BMI >30 kg/m2), will be placed on oral contraceptives for 2 months, then randomized into two intervention arms for an additional 2 months. At several key time points, synthetic steroid pharmacokinetics, gonadotropins (LH, FSH) and ovarian hormone levels (estradiol, progesterone), ovarian follicular activity by ultrasound monitoring, and cervical mucus testing will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-35
* BMI > 30kg/m2
* Proof of a normal breast and pelvic exam within last 9 months
* Self reported normal menstrual periods (24-35 days)
* Good general health
* In the investigator's opinion, are subject's veins suitable the repeat blood draws dictated by study protocol
* Single progesterone level during screening visit ≥ 3ng/mL
* Hematocrit ≥ 36%

Exclusion Criteria:

* Contradictions to COCs (history of deep vein thrombosis,myocardial infection, uncontrolled hypertension, pulmonary embolus, diabetes with vascular changes, stroke, migraines with neurologic changes, breast cancer, impaired liver function, uncontrolled thyroid disease, hypersensitivity or allergy to birth control)
* Smoker (must smoke 0 cigarettes)
* Actively seeking/involved in a weight loss program
* Currently pregnant/seeking pregnancy in the next 6 months
* Currently breast-feeding
* Past or current diagnosis of polycystic ovarian disease
* Recent use of birth control (Depot medroxyprogesterone: 6 months, Progestin implants: 6 months, Oral contraceptives, patch or ring: 2 months, Hormone impregnated IUD: 6 months)
* Currently taking medication that interferes with COC's (Rifampin, Carbamazepine, St. John's Wort)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2009-09; Primary Completion 2011-03 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Edelman, MD, MPH, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

REFERENCES:
- [Derived] Edelman AB, Cherala G, Munar MY, McInnis M, Stanczyk FZ, Jensen JT. Correcting oral contraceptive pharmacokinetic alterations due to obesity: a randomized controlled trial. Contraception. 2014 Nov;90(5):550-6. doi: 10.1016/j.contraception.2014.06.033. Epub 2014 Jun 27. PMID 25070547
- See also: (OHSU Women's Health Research Unit) — http://www.ohsuwomenshealth.com/research/index.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A prospective cohort study was conducted at the Oregon Health & Science University (OHSU) in Portland, OR, from March 2006 to September 2007. Recruitment included print ads in local newspapers, flyers posted in the Center for Women's Health & other OHSU clinics and public places, and electronic postings to web sites such as Craig's List.
Groups:
- All Participants: All participants were given a low dose oral contraceptive (Aviane) cyclically for 2 months
- Study Arm #1 (Aviane and Aviane): A very-low dose oral contraceptive given cyclically (21 days of active pills/cycle with a 7 day hormonal-free interval) for 2 cycles (56 days). A very-low dose oral contraceptive given continuously for 56 days (20mcg EE component, 28 days of active pills/cycle with no hormone free interval)
- Study Arm #2 (Aviane and Portia): A very-low dose oral contraceptive given cyclically (21 days of active pills/cycle with a 7 day hormonal-free interval) for 2 cycles (56 days). A low dose oral contraceptive given cyclically (30mcg EE component, 21 days of active pills/cycle with a 7 day hormonal-free interval) for two cycles
Period: Oral Contraceptives
Arm/Group | All Participants | Study Arm #1 (Aviane and Aviane) | Study Arm #2 (Aviane and Portia)
Started | 32 | 0 | 0
Completed | 31 | 0 | 0
Not Completed | 1 | 0 | 0
Period: Randomized Treatment
Arm/Group | All Participants | Study Arm #1 (Aviane and Aviane) | Study Arm #2 (Aviane and Portia)
Started | 0 | 17 | 15
Completed | 0 | 16 | 15
Not Completed | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Aviane and Aviane: A very-low dose oral contraceptive given cyclically (21 days of active pills/cycle with a 7 day hormonal-free interval) for 2 cycles (56 days). A very-low dose oral contraceptive given continuously for 56 days (20mcg EE component, 28 days of active pills/cycle with no hormone free interval)
- Aviane and Portia: A very-low dose oral contraceptive given cyclically (21 days of active pills/cycle with a 7 day hormonal-free interval) for 2 cycles (56 days). A low dose oral contraceptive given cyclically (30mcg EE component, 21 days of active pills/cycle with a 7 day hormonal-free interval) for two cycles
- Total: Total of all reporting groups
Arm/Group | Aviane and Aviane | Aviane and Portia | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 15 | 31
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (4) | 27 (4) | 29 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 31
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 15 | 31

OUTCOME MEASURES:

1. Primary Outcome: LNG Steady State at Baseline and Then Post-randomization
Description: The main goal is to test whether key pharmacokinetic parameters of levonordestrel (LNG) differ between obese women taking traditionally dosed OCs versus the interventional arms (i.e. using each obese subject as their own control).
Time Frame: baseline (2 months) and post-randomization (4 months)
Population: One subject discontinued prior to the completion of the baseline studies in the Aviane/Aviane arm
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Aviane & Aviane: A very-low dose oral contraceptive given cyclically (21 days of active pills/cycle with a 7 day hormonal-free interval) for 2 cycles (56 days). A very-low dose oral contraceptive given continuously for 56 days (20mcg EE component, 28 days of active pills/cycle with no hormone free interval)
- Aviane and Portia: A low dose oral contraceptive given cyclically (21 days of active pills/cycle with a 7 day hormonal-free interval) for 2 cycles (56 days). A low dose oral contraceptive given cyclically (30mcg EE component, 21 days of active pills/cycle with a 7 day hormonal-free interval) for two cycles
Arm/Group | Aviane & Aviane | Aviane and Portia
Number analyzed (Participants) | 16 | 15
ng/mL
  LNG steady state levels at baseline | 3.82 (1.28) | 3.13 (0.87)
  After randomization (4 months) | 3.01 (0.19) | 3.58 (0.35)

2. Secondary Outcome: LNG AUC
Description: Area under the curve post-randomization for levonorgestrel. AUC was calculated and extrapolated using post randomization in single daily samples drawn during Cycle 4 days 20-26. Serial repeat sampling to obtain a detailed PK curve was not performed to obtain this AUC. Subjects could provide samples during these days at times convenient to them and PK software accounted for the time between when the drug was dosed versus when the sample was drawn.
Time Frame: post-randomization (4 months)
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Aviane & Aviane | Aviane and Portia
Number analyzed (Participants) | 16 | 15
hr*ng/mL | 412 (255) | 283 (130)

3. Secondary Outcome: LNG AUC
Description: Baseline measurements of levonorgestrel AUC (on Aviane). Area under the curve at baseline for levonorgestrel. AUC was calculated from time zero to 168 hours and extrapolated to infinity from serial repeat sampling (0,0.5,1.1.5,2,3,4,6,8,12 hours and then single samples daily for 4 days between Cycles 1 and 2.
Time Frame: baseline (2 months)
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Aviane and Aviane | Aviane and Portia
Number analyzed (Participants) | 16 | 15
hr*ng/mL | 267 (115) | 199 (75)

4. Secondary Outcome: EE Steady State Baseline
Description: Steady state levels of ethinyl estradiol (EE) at baseline (2 months)
Time Frame: Baseline (2 months)
Population: One subject discontinued prior to the completion of the baseline cycle in the Aviane/Aviane arm
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Aviane & Aviane | Aviane and Portia
Number analyzed (Participants) | 16 | 15
ng/mL | 0.12 (0.04) | 0.1 (0.03)

5. Secondary Outcome: EE Steady State After Randomization
Description: Steady state levels of ethinyl estradiol (EE) post- randomization
Time Frame: Post-randomiziation 4 months
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Aviane & Aviane | Aviane and Portia
Number analyzed (Participants) | 16 | 15
ng/mL | 0.08 (0.08) | 0.11 (0.01)

ADVERSE EVENTS:
Arm/Group | Aviane and Aviane | Aviane and Portia
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 0/16 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes